CLINICAL TRIAL: NCT04830787
Title: Correlation Between Myocardial Deformation and Coronary Artery Morphology in Patients With Hypertrophic Cardiomyopathy and Analysis of Genetic Factors：A Prospective, Single-center, Case-control Study
Brief Title: Correlation Between Myocardial Deformation and Coronary Artery Tortuosity in Patients With Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TCAHCM
Record Dates: First submitted 2021-03-28; First posted 2021-04-05 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Myocardial Deformation; Coronary Artery Anomaly; Hypertrophic Cardiomyopathy; Genetic Mutation; Prognosis
Keywords: hypertrophic cardiomyopathy; tortuosity of coronary arteries; myocardial strain; prognosis; genetic mutation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertrophic cardiomyopathy: patients with hypertrophic cardiomyopathy
  Interventions: Other: no intervention
- control without hypertrophic cardiomyopathy: controls without hypertrophic cardiomyopathy

INTERVENTIONS:
Other: no intervention — there is no intervention, we just chose patients diagnosed with hypertrophic cardiomyopathy and underwent CAG, and patients without hypertrophic cardiomyopathy as control ,the two groups are matched with age, gender and hypertension.
  Groups: hypertrophic cardiomyopathy

SUMMARY:
Correlation between Myocardial Deformation and Coronary Tortuosity and Analysis of Genetic Factors Among Hypertrophic Cardiomyopathy Patients

DETAILED DESCRIPTION:
Excessive tortuosity of the coronary arteries (TCA) is a somewhat common finding in patients referred for coronary angiography, reported in 14-40% of patients referred for angiography. The presence of TCA has been associated with chest pain and myocardial perfusion abnormalities during stress in the absence of obstructive coronary artery disease. Fluid dynamic modeling suggests that stress-induced ischemia may be attributable to a reduction in distal coronary artery perfusion pressure from viscous and turbulence energy losses. The physiologic reasons for TCA are unclear. The roles of TCA on prognosis of HCM are also needed to explore. Pre-clinical studies where elastases and collagenases were used to alter arterial morphology together with genetic and pathologic analysis of rare clinical disorders such as arterial tortuosity syndrome have indicated that arterial tortuosity arises from abnormalities in arterial elastin fibers and extracellular matrix. Apart from inherited disorders, some but not all studies have linked TCA with hypertension and female sex, and with increased left ventricular (LV) mass from pressure but not volume overload and smaller heart size.

Hypertrophic cardiomyopathy (HCM) is associated with an increased left ventricular (LV) wall thickness. HCM is the most common genetic heart disease, characterized by marked clinical and morphologic heterogeneity. Diagnosis is usually based on the echocardiographic finding of unexplained left ventricular (LV) hypertrophy, defined by increased wall thickness in 1 or more LV segments. LV mass is generally assumed to be increased in patients with phenotypically expressed HCM, based largely on early pathological studies. TCA among HCM patients have not been studied. So, firstly, we choose HCM and non-HCM patients to investigate the relationship between TCA and HCM, and further explore the potential roles of TCA for prognosis in HCM.

In HCM patients, disruption of the ordered arrangement of myofibers alters normal cardiac mechanical function, resulting in temporal and spatial heterogeneity in regional myocardial contractility. Although global LV function is generally unaltered, asynchrony and asynergy in regional function lead to delayed diastolic relaxation and impaired diastolic filling. Whilst LV ejection fraction is frequently normal in both, LV strain assessment could differentiate, compared to normal person. Cardiovascular magnetic resonance (CMR), by virtue of its high-resolution volumetric reconstruction of the LV chamber, currently affords a highly accurate and reproducible quantitative assessment of mass . So secondly, we sought to establish if cardiovascular magnetic resonance myocardial feature tracking (CMR-FT), an emerging method allowing accurate assessment of myocardial deformation, differentiates between HCM with or without TCA. Additionally, we want to explore the potential genetic factor on TCA in HCM.

This is a single-center, retrospective, case control study that will evaluate the difference of TCA between HCM and non-HCM, and explore the prognostic roles of TCA in the first part. In the second part, we will use CMR-FT to compare the myocardial strain between HCM with or without TCA and analyze the relationship of strain and TCA. In the third part, we choose HCM patients and non-HCM to investigate potential genetic factors for TCA in HCM.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria to be eligible for participation in this study

  1. 18<age≤85；
  2. Patients with hypertrophic cardiomyopathy and without hypertrophic cardiomyopathy undergoing coronary angiography and echocardiography;
  3. Willing to sign informed consent.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study

  1. All coronary arteries can not be shown clearly in coronary angiography
  2. Prior coronary artery bypass surgery, valve prosthesis
  3. Connective tissue disease
  4. Cardiac dilatation(left ventricular end diastolic diameter, ≥55mm male，≥50mm female )
  5. Congenital heart failure, LVEF<35%
  6. Coronary total occlusion, changes in coronary morphology, such as long stents implantation（≥12mm）

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hypertrophic cardiomyopathy and without hypertrophic cardiomyopathy undergoing coronary angiography and echocardiography
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
coronary artery tortuosity and tortuosity score in hypertrophic cardiomyopathy patients | six months
  Severe tortuosity was defined as ≥2 consecutive curvatures of ≥180° in a major epicardial coronary artery ≥2 mm in diameter . Mild tortuosity was defined as either ≥3 consecutive curvatures of 45° to 90° in a major epicardial coronary artery, or ≥3 consecutive curvatures of 90° to 180° in an artery <2 mm in diameter. The tortuosity score was calculated as a sum of scores for each major epicardial coronary artery (left anterior descending, left circumflex, right coronary artery) with 0=no tortuosity, 1=mild tortuosity,2=tortuosity, 3=severe tortuosity. We will evaluate if the patients have coronary artery tortuosity and assess the number of tortuosity score for every coronary artery and add the score up for every patients.
prognostic roles of coronary artery tortuosity in hypertrophic cardiomyopathy | 2017/12/01-2022/07/01
  retrospectively included HCM patients with echocardiography and coronary angiography (CAG), in Fuwai Central China Cardiovascular Hospital from 1st Dec 2017 to 10th Jun 2021. All patients were followed up until the censoring day of 1st July 2022. The primary outcomes were composite of all-cause death, maglinant arrhythmia, ischemic stroke. Death was documented according to medical records, death certificates, or follow-up questionnaires by family members. Arrhythmia included ventricular fibrillation, sustained ventricular tachycardia, second-degree type II and third-degree atrioventricular block.
prognostic roles of coronary artery tortuosity in hypertrophic cardiomyopathy | 2017/12/01-2022/07/01
  etrospectively included HCM patients with echocardiography and coronary angiography (CAG), in Fuwai Central China Cardiovascular Hospital from 1st Dec 2017 to 10th Jun 2021. All patients were followed up until the censoring day of 1st July 2022. The secondary outcomes were composite of primary outcomes and rehospitalization.

SECONDARY OUTCOMES:
myocardial strain and strain rate in hypertrophic cardiomyopathy patients with coronary artery tortuosity | six months
  observe the difference of myocardial strain between hypertrophic cardiomyopathy with and without coronary artery tortuosity, Global longitudinal strain (GLS), global longitudinal strain rate (GLSR), global circumferential strain (GCS), global circumferential strain rate (GCSR), global radial strain (GRS), and global radial strain rate (GRSR) of the LV and RV will be calculated and segmental strain and strain rate will also be assessed respectively
genetic factors(such as genetic mutation site for HCM(MYBPC3,MYH7,ACTC1,TNNI3)) for hypertrophic cardiomyopathy patients with coronary artery tortuosity | two months
  do genetic testing, observe the difference for genetic factors such as gene mutation for hypertrophic cardiomyopathy with and without coronary artery tortuosity, all the 40 genes which has been found to be implicated in HCM will be tested, such as MYBPC3, MYH7, TPM1,TNNT2 and TNNI3.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Ge, PhD, Study Chair — Henan Provincial People's Hospital; You Zhang, PhD, Study Director — Henan Provincial People's Hospital; Shan Wang, MD, Study Director — Henan Provincial People's Hospital; Yi Huang, MD, Study Director — Henan Provincial People's Hospital; Qing Lin, MD, Study Director — Henan Provincial People's Hospital; Yabing Li, MD, Study Director — Henan Provincial People's Hospital; Lei Yu, MD, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Central China Fuwai Hospital, Heart Center of Henan Provincal People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
It will be decided by patients , hospital and Chinese health authority.

REFERENCES:
- [Background] Li Y, Shen C, Ji Y, Feng Y, Ma G, Liu N. Clinical implication of coronary tortuosity in patients with coronary artery disease. PLoS One. 2011;6(8):e24232. doi: 10.1371/journal.pone.0024232. Epub 2011 Aug 31. PMID 21904618
- [Background] Eleid MF, Guddeti RR, Tweet MS, Lerman A, Singh M, Best PJ, Vrtiska TJ, Prasad M, Rihal CS, Hayes SN, Gulati R. Coronary artery tortuosity in spontaneous coronary artery dissection: angiographic characteristics and clinical implications. Circ Cardiovasc Interv. 2014 Oct;7(5):656-62. doi: 10.1161/CIRCINTERVENTIONS.114.001676. Epub 2014 Aug 19. PMID 25138034
- [Background] Barilla F, Romeo F, Rosano GM, Valente A, Reale A. Coronary artery loops and myocardial ischemia. Am Heart J. 1991 Jul;122(1 Pt 1):225-6. doi: 10.1016/0002-8703(91)90781-c. No abstract available. PMID 2063741
- [Background] Vorobtsova N, Chiastra C, Stremler MA, Sane DC, Migliavacca F, Vlachos P. Effects of Vessel Tortuosity on Coronary Hemodynamics: An Idealized and Patient-Specific Computational Study. Ann Biomed Eng. 2016 Jul;44(7):2228-39. doi: 10.1007/s10439-015-1492-3. Epub 2015 Oct 23. PMID 26498931
- [Background] Maron BJ, McKenna WJ, Danielson GK, Kappenberger LJ, Kuhn HJ, Seidman CE, Shah PM, Spencer WH 3rd, Spirito P, Ten Cate FJ, Wigle ED; Task Force on Clinical Expert Consensus Documents. American College of Cardiology; Committee for Practice Guidelines. European Society of Cardiology. American College of Cardiology/European Society of Cardiology clinical expert consensus document on hypertrophic cardiomyopathy. A report of the American College of Cardiology Foundation Task Force on Clinical Expert Consensus Documents and the European Society of Cardiology Committee for Practice Guidelines. J Am Coll Cardiol. 2003 Nov 5;42(9):1687-713. doi: 10.1016/s0735-1097(03)00941-0. No abstract available. PMID 14607462
- [Background] Weidemann F, Mertens L, Gewillig M, Sutherland GR. Quantitation of localized abnormal deformation in asymmetric nonobstructive hypertrophic cardiomyopathy: a velocity, strain rate, and strain Doppler myocardial imaging study. Pediatr Cardiol. 2001 Nov-Dec;22(6):534-7. doi: 10.1007/s002460010293. Epub 2001 Dec 4. PMID 11894166
- [Background] Salton CJ, Chuang ML, O'Donnell CJ, Kupka MJ, Larson MG, Kissinger KV, Edelman RR, Levy D, Manning WJ. Gender differences and normal left ventricular anatomy in an adult population free of hypertension. A cardiovascular magnetic resonance study of the Framingham Heart Study Offspring cohort. J Am Coll Cardiol. 2002 Mar 20;39(6):1055-60. doi: 10.1016/s0735-1097(02)01712-6. PMID 11897450